CLINICAL TRIAL: NCT05008029
Title: Cast Immobilization Without Reduction vs. Reduction Under General Anesthesia in Metaphyseal Fractures of the Distal Radius.
Brief Title: Immobilization Without Reduction vs. Reduction Under General Anesthesia in Metaphyseal Fractures of the Distal Radius
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment time ended, but sample size was not completed.
Sponsor: Instituto de Ortopedia Infantil Roosevelt (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021012101
Record Dates: First submitted 2021-06-10; First posted 2021-08-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Radius Fracture Distal
Keywords: radius fracture; children; conservative treatment; distal radius
MeSH Terms: conditions — Wrist Fractures; Radius Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will analyze the database without knowing which treatment arm each participant was allocated. He does not work in the center where the study will be carried out, nor does he contact the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In situ immobilization (Experimental): Immobilization without reducing the radius fracture and above-elbow casting.
  Interventions: Procedure: In situ immobilization
- Reduction under general anesthesia (Active Comparator): Radius closed reduction under general anesthesia and above-elbow casting. Percutaneous fixation with K-wires, a sugar tong splint immobilization, and a nerve block if needed.
  Interventions: Procedure: Reduction under general anesthesia

INTERVENTIONS:
Procedure: In situ immobilization — Immobilization with an above-elbow cast. A 2, 3, or 4-year orthopedic resident or pediatric orthopedic fellow supervised by a pediatric orthopedic surgeon will perform the procedure without reduction, sedation, or anesthesia. Analgesia will be administered with paracetamol at doses of 10-15 mg/kg/dose or tramadol 0.5-1mg/kg/dose. Supposing immobilization is not satisfactory, or the patient or family member does not authorize the procedure to be carried out by staff in training. In that case, the procedure will be supported or carried out by the pediatric orthopedic surgeon.
  Arms: In situ immobilization
Procedure: Reduction under general anesthesia — The participants will receive paracetamol at 10-15 mg/kg/dose or tramadol 0.5-1 mg/kg/dose for pain control until the time of surgery. Under general anesthesia, radius closed reduction, and above-elbow casting will be performed. After the reduction maneuvers, the radius reduction is satisfactory if the translation in the coronal and sagittal planes of less than 50% and angulation in the same planes is less than 10 °. If the radius does not remain reduced, it is unstable. Unstable fractures require percutaneous fixation with K-wires, a sugar tong splint immobilization, and a nerve block. The procedures will be carried out by a 2, 3, or 4-year orthopedic resident or pediatric orthopedic fellow under the supervision of a child orthopedist. Suppose reduction is not satisfactory or the patient or parent doesn´t authorize the procedure performed by personnel in training. In that case, the procedure will be supported or carried out by the pediatric orthopedic surgeon.
  Arms: Reduction under general anesthesia

SUMMARY:
Distal radius metaphyseal fractures are the most frequent in the pediatric population. The current treatment for angulated or shortened fractures is effective. Still, it exposes children to anesthetic risks supported by the pain generated by the reduction. Due to the excellent remodeling capacity of bone at an early age, it is questionable whether an anatomical reduction is necessary.

The clinical experiment's objective is to compare the functional result of immobilization without reducing angulated or displaced metaphyseal fractures of the distal radius against fractures brought to reduction under general anesthesia. Means difference in function subdomain of the upper limb of the PROMIS® scale is the primary outcome. The secondary results are wrist mobility, radius alignment, wrist articular relationships, and surgical complications.

DETAILED DESCRIPTION:
The participant will be recruited in one center. If participants and their parents accept to participate in this study, treatments will be randomly allocated using the Big Stick Design technique with a maximum tolerated imbalance of 2. The sequence will be generated by a research assistant who is completely independent of the study, does not know the purpose of the study and the interventions. Each of the random numbers will be stored in an opaque envelope sealed externally with the order in which they should be opened.

Patient registration and follow-up information will be stored in REDCap®. Clinical and radiographic outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children from 5 years to 10 years
* Unilateral metaphyseal distal radius fracture
* Fracture shortening of 0 to 10mm or angulation of 10 ° to 20 ° in the oblique plane. (AO 23-M 2-3 or 23r-M 2-3)
* Admission in the first 14 days after the fracture

Exclusion Criteria:

* Polytrauma: Injury Severity Score (ISS)> 16
* Associated fracture in the same limb.
* Neuromuscular pathology (e.g., cerebral palsy, spinal muscular atrophy, Duchenne disease)
* Open fractures.
* History of fractures, septic arthritis, or osteomyelitis in the same limb.
* Neurological or vascular injury in the fractured upper limb.
* Known alteration of bone metabolism (e.g., osteogenesis imperfecta, rickets, osteopetrosis, skeletal dysplasias, lysosomal storage diseases).
* Congenital longitudinal deficiency.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Upper limb function | 6 months
  Assess upper extremity function with PROMIS Physical Function, Upper Extremity subdomain. The investigators will apply the parent-proxy version between 5 and 7 years old and the pediatric version between 8 and 10.

SECONDARY OUTCOMES:
Wrist range of motion | 3 and 6 months
  Wrist passive degrees of flexion and extension measured with a goniometer aligned with the forearm axis and the second metacarpal.
  Pronation and supination. The investigators will ask the patient to hold a pencil vertically with the ulnar edge of the forearm on the table and the elbow flexed 90 °. The wrist is rotated medially or laterally, respectively. One arm of the goniometer is placed on the table and the other is aligned with the pencil, the degrees obtained must be subtracted from 90 °.
Ulnar variance | 9 months
  The investigators will consider the ulnar variance as the distance between the most distal aspect of the metaphysis of the radius and the ulna according to the Hafner distal-distal method (DIDI).
Deformity | 2 weeks, 3 months and 9 months
  Angulation in the oblique plane

OTHER OUTCOMES:
Number of patients with anesthetic complications | During and immediately after the intervention
  Number of participants with one of the following complications: Rash, pruritus, nausea, vomiting, bruising. hallucinations, toxicity, neurological injury, seizures, respiratory depression, bronchospasm, laryngospasm, cardiovascular events, malignant hyperthermia, and death.
Presence of a pressure ulcer (NPUAP scale) | 2 and 6 weeks
  Pressure zones caused by plaster and classified with the National Pressure Ulcer Advisory Panel scale. The score range from 1 to 4. Higher scores mean a worse outcome. Unclassifiable lesions or those with deep tissue lesions will be reclassified to type 3 or 4 lesions after surgical debridement. For the purposes of the study, the value of the reclassification will be taken.
Patients's pain control | 2 and 6 weeks
  Days of analgesic consumption
Number of patients with pin tract infection (Dahl scale) | 2 and 6 weeks
  Only in patients with percutaneous fixation with K-wires will the pin tract infection be classified with the Dahl scale.
Number of patients with reintervention | 0 to 9 months
  Surgical intervention in the fractured radius during the nine months after the assigned treatment due to nonunion, re-displacement, or malunion

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Garcia, MD, Principal Investigator — Instituto Roosevelt
Locations (1):
- Instituto Roosevelt, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Study information will be available through the institutional website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: On permission request
URL: https://www.institutoroosevelt.com

REFERENCES:
- [Background] Marson BA, Ng JWG, Craxford S, Chell J, Lawniczak D, Price KR, Ollivere BJ, Hunter JB. Treatment of completely displaced distal radial fractures with a straight plaster or manipulation under anaesthesia. Bone Joint J. 2021 May;103-B(5):902-907. doi: 10.1302/0301-620X.103B.BJJ-2020-1740.R1. Epub 2021 Mar 12. PMID 33709769
- [Derived] Garcia-Rueda MF, Bohorquez-Penaranda AP, Gil-Laverde JFA, Aguilar-Sierra FJ, Mendoza-Pulido C. Casting Without Reduction Versus Closed Reduction With or Without Fixation in the Treatment of Distal Radius Fractures in Children: Protocol for a Randomized Noninferiority Trial. JMIR Res Protoc. 2022 Apr 14;11(4):e34576. doi: 10.2196/34576. PMID 35436224

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT05008029/Prot_SAP_000.pdf